CLINICAL TRIAL: NCT06476119
Title: OPTImaL:Optimisation of Treatment for Patients With Low Stage Triple-negative Breast Cancer With High Stromal Tumor-infiltrating Lymphocytes
Acronym: OPTImaL
Status: Recruiting | Type: Observational
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Maarten van de Weijden Foundation (Unknown); AVL Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: M24OTI
Record Dates: First submitted 2024-06-07; First posted 2024-06-26 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer Stage I; Triple Negative Breast Cancer (TNBC)
Keywords: High (stromal Tumor-Infiltrating-Lymphocytes) sTIL score
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Chemotherapy, Adjuvant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — ctDNA samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Optimisation cohort: patients will be treated with surgery and adjuvant radiotherapy following local/national guidelines, while chemotherapy will be omitted
  Interventions: Other: No adjuvant chemotherapy
- Control cohort: patients will be treated with surgery, adjuvant radiotherapy and adjuvant chemotherapy following local/national guidelines
  Interventions: Drug: Adjuvant chemotherapy

INTERVENTIONS:
Drug: Adjuvant chemotherapy — adjuvant chemotherapy according to local/ national guidelines
  Other Names: according to local/ national guidelines
  Groups: Control cohort
Other: No adjuvant chemotherapy — no adjuvant chemotherapy
  Groups: Optimisation cohort

SUMMARY:
The aim of this study is to investigate whether subjects with breast cancer that have certain favorable features, after performing the surgery and radiation, the chemotherapy can be safely omitted in the treatment. In addition, the investigation looks at whether the omission of chemotherapy ensures a better quality of life. Participants decide, in consultation with their treating physician, whether they choose to be treated with adjuvant chemotherapy or not.

ELIGIBILITY:
Inclusion Criteria:

* Female or male patients;
* >=18 years;
* Written informed consent;
* TNBC (defined as: invasive carcinoma; ER/PR expression 0-9%; Human Epidermal Growth Factor Receptor 2 [HER2] negative [0, 1+ or 2+ on immunohistochemistry, without HER2 amplification on in-situ hybridization]) on the diagnostic biopsy and the surgical specimen;
* Pathological stage I TNBC (according to the TNM staging 8th edition):

  * pT1a/b/c (≤2 cm), confirmed by an invasive component of ≤2 cm on the surgical specimen (microinvasive disease [pT1mi, ≤1 mm) is not allowed);
  * pN0, confirmed by absence of malignant cells in the sentinel lymph node or any other lymph node after surgery (isolated tumor cells [N0(i+)] are not allowed);
* No evidence of nodal or distant metastases (cN0M0) on pre and/or postoperative imaging examinations (performed following local/national guidelines, but must include an 18F-fluorodeoxyglucose positron emission tomography/computed tomography [18F-FDG-PET/CT, at least from skull base to upper legs] or computed tomography [CT] of neck/chest/abdomen/pelvis [CT only if 18F-FDG-PET/CT would not be available; 18F-FDG-PET/CT mandatory in the Netherlands]);
* sTIL score of ≥50% for patients ≥40 years at the time of TNBC diagnosis and ≥75% for patients <40 years at the time of TNBC diagnosis on an H&E FFPE tissue slide on the surgical specimen, according to International Immuno-Oncology Biomarker Working Group on Breast Cancer (formerly International TILs Working Group) guidelines, by local and central review
* Has undergone curative breast surgery (breast-conserving surgery or mastectomy and surgical axillary staging [including at least sentinel lymph node procedure]);
* Absence of recurrence between curative breast surgery and expression of patient preference;
* Eligible for radiotherapy (if indicated).

Exclusion Criteria:

* Prior disease history of invasive and/or non-invasive breast cancer, or ongoing treatment for invasive and/or non-invasive breast cancer;
* Multifocal, multicentric or bilateral breast cancer at the time of screening;
* Administration of neoadjuvant systemic therapy;
* Presence of lymphovascular invasion on the diagnostic biopsy and/or the surgical specimen;
* Other invasive malignancy within 5 years prior to inclusion, with the exception of ade-quately treated non-melanoma skin cancer, localized cervical cancer, localized and Gleason ≤6 prostate cancer;
* Uncontrolled severe illness or medical condition;
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be assessed and discussed with the patient before the enrolment in the in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with pathological stage I TNBC (pT1a/b/cN0) and a high sTIL score (defined as ≥50% for patients ≥40 years; ≥75% for patients <40 years)
Sampling Method: Probability Sample
Enrollment: 490 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2032-09-15 (Estimated); Study Completion 2034-09-15 (Estimated)

PRIMARY OUTCOMES:
Disease recurrence Free Interval (DRFI) - optimalisation cohort per-protocol population | up to 96 months after inclusion of the last patient
  Number of patients with distant recurrence or death in per-protocol population of the optimisation cohort

SECONDARY OUTCOMES:
Disease recurrence Free Interval (DRFI) - optimalisation cohort intention to treat population | up to 96 months after inclusion of the last patient
  Number of patients with distant recurrence or death in intention to treat population of the optimisation cohort
Disease recurrence Free Interval (DRFI) - control cohort | up to 96 months after inclusion of the last patient
  Number of patients with distant recurrence or death in control cohort
Invasive disease-free survival (IDFS) - optimalisation cohort per-protocol population | up to 96 months after inclusion of the last patient
  Number of patients with breast tumor recurrence or death in the per-protocol population of the optimisation cohort
Invasive disease-free survival (IDFS) - optimalisation cohort intention-to-treat population | up to 96 months after inclusion of the last patient
  Number of patients with breast tumor recurrence or death in the the intention-to-treat population of the optimisation cohort
Invasive disease-free survival (IDFS) - control cohort | up to 96 months after inclusion of the last patient
  Number of patients with breast tumor recurrence or death in the control cohort
disease recurrence free survival (DRFS) - optimalisation cohort per-protocol population | up to 96 months after inclusion of the last patient
  time between inclusion and first distant recurrence or death from any cause in the per-protocol population of the optimisation cohort
disease recurrence free survival (DRFS) - optimalisation cohort the intention-to-treat population | up to 96 months after inclusion of the last patient
  time between inclusion and first distant recurrence or death from any cause in the intention-to-treat population of the optimisation cohort population of the optimisation cohort
disease recurrence free survival (DRFS) - control cohort | up to 96 months after inclusion of the last patient
  time between inclusion and first distant recurrence or death from any cause in the control cohort
Recurrence-free survival (RFS) - optimalisation cohort per-protocol population | up to 96 months after inclusion of the last patient
  time between inclusion and invasive ipsilateral breast tumor recurrence, local-regional invasive recurrence, distant recurrence or death from any cause in the per-protocol population of the optimisation cohort;
Recurrence-free survival (RFS) - optimalisation cohort the intention-to-treat population | up to 96 months after inclusion of the last patient
  time between inclusion and invasive ipsilateral breast tumor recurrence, local-regional invasive recurrence, distant recurrence or death from any cause in the the intention-to-treat population of the optimisation cohort;
Recurrence-free survival (RFS) - control cohort | up to 96 months after inclusion of the last patient
  time between inclusion and invasive ipsilateral breast tumor recurrence, local-regional invasive recurrence, distant recurrence or death from any cause in the control cohort;
Overal Survival (OS) - optimalisation cohort per-protocol population | up to 96 months after inclusion of the last patient
  time between inclusion and death from any cause in the per-protocol population of the optimisation cohort;
Overal Survival (OS) - optimalisation cohort intention-to-treat population | up to 96 months after inclusion of the last patient
  time between inclusion and death from any cause in the the intention-to-treat population of the optimisation cohort;
Overal Survival (OS) - control cohort | up to 96 months after inclusion of the last patient
  time between inclusion and death from any cause in the control cohort;
Health related Quality of Life (HRQoL) - (European Organisation on Research and Treatment of Cancer) EORTC questionnaire QLQ-C30 | up to 2 years after inclusion
  Difference in QoL assessed with the EORTC QLQ-C30 questionnaires between the optimisation and the control group. A higher score indicates a higher symptom burden.
Health related Quality of Life (HRQoL) - (European Organisation on Research and Treatment of Cancer) EORTC questionnaire QLQ-BR45 | up to 2 years after inclusion
  Difference in QoL assessed with the EORTC QLQ-BR45 questionnaires between the optimisation and the control group. A higher score indicates a higher symptom burden.
Fear of recurrence | up to 2 years after inclusion
  Assessed with questionnaires to determine the difference in optimisation and control group
Worries about health | up to 2 years after inclusion
  Assessed with questionnaires to determine the difference in optimisation and control group. A higher score indicates a higher symptom burden.
Cost effectiveness measured by quality-adjusted-life years (QALYs) | up to 2 years after inclusion
  Measured per Quality-Adjusted Life Years (QALYs)
Cost effectiveness measured per incremental cost-effectiveness ratio (ICER) | up to 2 years after inclusion
  Measured per incremental cost-effectiveness ratio (ICER)

CONTACTS AND LOCATIONS:
Overall Officials: Marleen Kok, MD, Principal Investigator — Antoni van Leeuwenhoek
Locations (28):
- Netherlands (28):
  - Zuyderland Medisch Centrum, Sittard-Geleen, Limburg
  - Medical spectrum Twente, Enschede, Overijssel
  - Noordwest Ziekenhuisgroep, Alkmaar
  - Flevoziekenhuis, Almere Stad
  - Meander Medisch Centrum, Amersfoort
  - Antoni van Leeuwenhoek, Amsterdam
  - Onze Lieve Vrouwe Gasthuis (OLVG), Amsterdam
  - Rijnstate, Arnhem
  - Amphia ziekenhuis, Breda
  - Deventer Ziekenhuis, Deventer
  - Ziekenhuis Gelderse Vallei, Ede
  - Catharina Ziekenhuis, Eindhoven
  - Jeroen Bosch ziekenhuis, Eindhoven
  - St. Jansdal, Harderwijk
  - Ziekenhuisgroep Twente, Hengelo
  - Tergooi ziekenhuizen, Hilversum
  - Spaarne Gasthuis, Hoofddorp
  - Dijklander ziekenhuis, Hoorn
  - MCL, Leeuwarden
  - LUMC, Leiden
  - MUMC, Maastricht
  - St. Antonius ziekenhuis, Nieuwegein
  - Radboud UMC, Nijmegen
  - Erasmus Medical Center Cancer Institute, Rotterdam
  - Franciscus Gasthuis & Vlietland, Schiedam
  - Haaglanden Medisch Centrum, The Hague
  - VieCuri Medisch Centrum voor Noord-Limburg, Venlo
  - Isala, Zwolle

IPD SHARING:
Plan to Share IPD: No
no IPD plan